CLINICAL TRIAL: NCT01060345
Title: A Pilot Study of Chemo-prevention of Green Tea in Women With Ductal Carcinoma in Situ (DCIS)
Brief Title: A Pilot Study of Chemo-prevention of Green Tea in Women With Ductal Carcinoma in Situ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug no longer available
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 09-151-B
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Results first posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-03

CONDITIONS: Ductal Carcinoma in Situ
Keywords: DCIS
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating | interventions — polyphenon E; Tea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Women with Ductal Carcinoma in Situ (Experimental): Women who have been diagnosed with ductal carcinoma in situ (DCIS) and will be taking Polyphenon E
  Interventions: Drug: Polyphenon E

INTERVENTIONS:
Drug: Polyphenon E — three 200mg capsules (600mg total dose of the study drug) with food (within one hour of eating a substantial meal) daily for a minimum of 4 weeks, or until the day before surgery
  Other Names: Green tea

SUMMARY:
The purpose of this study is to find molecular signs (biomarkers) to better understand the role of green tea as an anti-cancer and anti-inflammation agent in women with newly-diagnosed ductal carcinoma in situ (DCIS).

DETAILED DESCRIPTION:
Many studies have shown that green tea may have anti-cancer and anti-inflammatory effects in cancer cells and animal models of breast cancer. Some studies have found that Asian women who drink many cups of green tea have lower rates of breast cancer. Green tea may have an effect on proliferative and inflammatory pathways. Women with ductal carcinoma in situ (DCIS) have been found to have inflammation in the breast tissue surrounding DCIS lesions. Inflammatory pathways are being studied for a possible link to cancer. This study is designed to evaluate changes in biomarkers of proliferation, inflammation, and angiogenesis in response to green tea intake.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DCIS by breast core biopsy with a corresponding lesion on breast MRI of at least 1-cm3 in volume.
* Patients may have undergone treatment with prior chemotherapy if this was greater than 12 months prior to current diagnosis.
* Age >18 years.
* ECOG performance status <2 (Karnofsky >60%)
* Life expectancy of greater than 12 months.
* Normal organ and marrow function as defined below:
* leukocytes >3,000/mcL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* total bilirubin within normal institutional limits
* AST(SGOT) & ALT(SGPT)within normal institutional limits
* creatinine <1.5 times institutional upper limit of normal or creatinine clearance >60 mL/min/1.73 m2
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnancy
* Patients who have undergone prior excisional biopsy for DCIS.
* Patients who are unable to undergo MRI due to claustrophobia or other reason.
* Patients with ipsilateral treatment for DCIS or breast cancer within 12 months prior to entering this study.
* Patients receiving any other chemotherapy or investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to green tea extracts or sensitivity to green tea.
* Uncontrolled concurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nora Jaskowiak, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Women With Ductal Carcinoma in Situ
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 56.8 [43 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in K167 Staining
Time Frame: Prior to starting study and after 4-6 weeks of treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

2. Secondary Outcome: Decrease in MRI Volume and Signal Enhancement Ratio (SER) of the Breast Lesion From Pre- to Post-treatment.
Time Frame: Prior to study start and 4-6 weeks after treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Percent Staining of CD68 in Breast Tissue
Time Frame: Prior to study start and 4-6 weeks after treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Percent Staining of CD31 in Breast Tissue
Time Frame: Prior to study start and 4-6 weeks after treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Percent Staining of VEGF in Breast Tissue
Time Frame: Prior to study start and after 4-6 weeks of treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in Serum Levels of IGF-1
Time Frame: Prior to study start and after 4-6 weeks of treatment
Population: 0 analyzed, data not collected as the study stopped early due to lack of drug supply
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety of Green Tea Ingestion
Description: Number of patients with adverse event.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Women With Ductal Carcinoma in Situ
Number analyzed (Participants) | 20
Participants | 6

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Women With Ductal Carcinoma in Situ
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 6/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Women With Ductal Carcinoma in Situ (N=20)
Fatigue (General disorders) | 1
Anxiety (Psychiatric disorders) | 2
Headache (Nervous system disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Palpitations (Cardiac disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes